CLINICAL TRIAL: NCT03885349
Title: Motivational Strategies in Batterer Intervention Programs for Intimate Partner Violence Offenders With Alcohol/Drug Abuse Problems: An Experimental Study
Brief Title: Motivational Strategies in Batterer Intervention Programs for Offenders With Alcohol/Drug Abuse Problems (IMP-ADAPs)
Acronym: IMP-ADAPs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Collaborators: Ministerio de Sanidad, Servicios Sociales e Igualdad (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H1537520365110
Record Dates: First submitted 2019-02-05; First posted 2019-03-21 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Intimate Partner Violence Against Women; Alcohol Abuse; Drug Abuse
Keywords: Intimate partner violence; Alcohol; Drug; Batterer intervention programs
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBIP+ ADAPs-IMP (Experimental): Experimental condition: Standard batterer intervention program (SBIP) plus individualized motivational plan (IMP) focused in alcohol and/or drugs abuse problems (ADAPs).
  Interventions: Behavioral: SBIP+ ADAPs-IMP
- SBIP+IMP (Active Comparator): Control condition: Standard batterer intervention program plus individualized motivational plan (SBIP+IMP)
  Interventions: Behavioral: SBIP+IMP

INTERVENTIONS:
Behavioral: SBIP+ ADAPs-IMP — Standard batterer intervention program plus Individualized Motivational Plans adapted to alcohol and/or drug abuse problems. The SBIP consist of 70 hr of a cognitive-behavioral intervention including discussion topics such as sexism, sex roles, and gender equality. The intervention phase consisted of six modules in which different intervention techniques were applied (i.e., group dynamics, roleplaying, videos, training in cognitive restructuring, emotion management skills). The IMP included a set of motivational strategies to increase treatment compliance and motivation for change and had four main strategies: (a) five individual motivational interviews, to identify IPV related personal goals and follow up their achievement (in this case, one of the goals has to be related to ADAPs); (b) three group sessions where participants share their goals; (c) therapists follow-up and reinforcement of participants' goals; and (d) use of retention techniques.
  Arms: SBIP+ ADAPs-IMP
Behavioral: SBIP+IMP — Standard batterer intervention program plus Individualized Motivational Plans. The SBIP consist of 70 hr of a cognitive-behavioral intervention including discussion topics such as sexism, sex roles, and gender equality. The intervention phase consist of six modules in which different intervention techniques are applied (i.e., group dynamics, roleplaying, videos, training in cognitive restructuring, emotion management skills). The IMP include a set of motivational strategies to increase treatment compliance and motivation for change and has four main strategies: (a) five individual motivational interviews, to identify IPV related personal goals and follow up their achievement; (b) three group sessions where participants share their goals, explain their progress to the group, and receive feedback, support and advice from the group; (c) therapists follow-up and reinforcement of participants' goals; and (d) use of retention techniques.
  Arms: SBIP+IMP

SUMMARY:
Alcohol and/or drug abuse problems (ADAPs) have been consistently identified in the scientific literature as a risk factor of intimate partner violence against women (IPVAW). Around 50% of IPVAW offenders referred to batterer intervention programs (BIPs) have ADAPs. ADAPs are also one of the main predictors of BIPs dropout. In Spain, the majority of BIPs do not fit the intervention to specific needs or characteristics of IPVAW offenders, such as those with ADAPs. The aim of this research is to assess the effectiveness of a new motivational strategy adapted to IPVAW offenders with ADAPs, aiming to increase treatment adherence and to improve BIPs outcomes. The motivational strategy will include an individualized motivational plan (IMP) developed for each participant with ADAPs (IMP-ADAPs). In these IMPs one of the main aims will be to reduce alcohol and/or drug consumption. The current study will use a randomized control trial. Participants with ADAPs will be allocated to one of two treatment conditions: experimental condition: Standard batterer intervention program (SBIP) plus individualized motivational plan focused in ADAPs (SBIP+ ADAPs-IMP), and control condition: Standard batterer intervention program plus individualized motivational plan (SBIP+IMP). Primary/final outcomes will be recidivism and ADAPs reduction. Secondary/proximal outcomes will include treatment adherence related variables, violence related attitudes and attributions, self-control and psychological adjustment. Outcome variables will be assessed at baseline, at the end of the intervention, and at six months after the intervention will be finished.

ELIGIBILITY:
Inclusion Criteria:

* Males convicted of IPV against their partner or ex-partner
* Alcohol and/or drugs abuse problems

Exclusion Criteria:

* No current severe psychological disorders

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2019-03-04 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in alcohol abuse problems | At baseline, at 12 months (end of intervention), and at 18 months (follow-up)
  Alcohol Use Disorders Identification Test. Saunders, Aasland, Babor, De la Fuente, & Grant, 1993. Total scale range: 0-20 (Higher values indicate worse outcome).
Change in cannabis abuse problems | At baseline, at 12 months (end of intervention), and at 18 months (follow-up)
  Severity Dependence Scale. Gossop et al., 1995. Total scale range: 0-15 (Higher values indicate worse outcome).
Change in cocaine abuse problems | At baseline, at 12 months (end of intervention), and at 18 months (follow-up)
  Severity Dependence Scale. Gossop et al., 1995. Total scale range: 0-15 (Higher values indicate worse outcome).
Change in self-reported physical intimate partner violence against women | At baseline, at 12 months (end of intervention), and at 18 months (follow-up)
  Self-reported physical violence sub-scale from the Conflict Tacticts Scale. Straus, Hamby, Boney-McCoy y Sugarman, 1996. Total scale range: 0-72 (Higher values indicate worse outcome).
Change in self-reported psychological intimate partner violence against women | At baseline, at 12 months (end of intervention), and at 18 months (follow-up)
  Self-reported psychological violence sub-scale from the Conflict Tacticts Scale. Straus, Hamby, Boney-McCoy y Sugarman, 1996. Total scale range: 0-72 (Higher values indicate worse outcome).
Change in risk of recidivism | At baseline, at 12 months (end of intervention), and at 18 months (follow-up)
  The Spousal Assault Risk Assessment. SARA; Kropp y Hart, 2000. Total scale range: 0-40 (Higher values indicate worse outcome)
Police-reported recidivism | At 18 months (follow-up)
  Ministry of Home Affairs' monitoring system for IPV. This system includes information on further incidents of violence by individuals convicted of IPV and reported by any of the institutions involved in victim protection services. Recidivism will be considered to have occurred when this information appear in the system in the 6 months after completing the intervention.

SECONDARY OUTCOMES:
Therapeutic alliance | 4 weeks after the first session of the intervention
  Working Alliance Inventory Shortened Observer-rated version (WAI-O-S; Tichenor & Hill, 1989). Total scale range: 0-74 (Higher values indicate better outcome)
Change in motivation | At baseline, at 6 months, and at 12 months (end of intervention)
  Based on the transtheoretical model of change (Prochaska and DiClemente, 1982; Prochaska et al., 1992), therapists will rate participants' stage of change (pre-contemplation, contemplation, preparation, action, and maintenance). Total range: 1-5 (Higher values indicate better outcome).
Change in impulsivity | At baseline and at 12 months (end of intervention)
  Plutchik Impulsivity Scale; Plutchnik y Van Pragg, 1989. Total scale range: 11-44 (Higher values indicate worse outcome)
Change in depressive symptomatology | At baseline and at 12 months (end of intervention)
  Spanish reduced version of the Center for Epidemiology Studies-Depression Scale; Herrero y Gracia, 2007. Total scale range: 7-28 (Higher values indicate worse outcome)
Change in self-esteem | At baseline and at 12 months (end of intervention)
  Rosenberg Self-Esteem Scale. Rosenberg, 1965. Total scale range: 10-40 (Higher values indicate better outcome)
Attributions of Responsibility | At baseline and at 12 months (end of intervention)
  Intimate Partner Violence Responsibility Atribution Scale. Lila, Oliver, Catalá-Miñana, Galiana y Gracia, 2014. Three sub-scales: responsibility attribution to the legal system (sub-scale range: 4-20), responsibility attribution to the victim (sub-scale range: 4-20), and responsibility attribution to the offender personal context (sub-scale range: 4-20). Higher values indicate worse outcome.
Change in perceived severity of intimate partner violence against women | At baseline and at 12 months (end of intervention)
  Severity Perception of Intimate Partner Violence Against Women Scale. Gracia, García y Lila (2011). Total scale range: 8-80 (Higher values indicate better outcome)
Change in acceptability of intimate partner violence against women | At baseline and at 12 months (end of intervention)
  Acceptability of Intimate Partner Violence Against Women Scale. Martín-Fernández, Gracia, Marco, Vargas, Santirso and Lila (2018). Total scale range: 0-40 (Higher values indicate worse outcome)
Change in benevolent sexism | At baseline and at 12 months (end of intervention)
  Ambivalent Sexism Inventory. Glick y Fiske, 1996. Two sub-scales: Benevolent sexism (sub-scale range: 0-55) and Hostile sexism (sub-scale range: 0-55). Higher values indicate worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Marisol Lila, PhD, Principal Investigator — University of Valencia
Locations (1):
- Faculty of Psychology, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No